CLINICAL TRIAL: NCT01583556
Title: Optional Follow-up Visits for Common, Low-risk Arm Fractures
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, David C. Ring, MD, Director of Research, Hand Service, Massachusetts General Hospital
Other Study IDs: 2012P000632
Record Dates: First submitted 2012-03-27; First posted 2012-04-24 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Mallet Fracture; Metacarpal Fracture; Metacarpal Neck Fracture; Distal Radius Fracture; Radial Head Fracture
Keywords: Adult; English speaking; Fractures; Excellent prognosis; Upper Extremity
MeSH Terms: conditions — Wrist Fractures; Radial Head and Neck Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard treatment: This study will employ a prospective, non-randomized design. After the questionnaires are filled the patients choose whether or not to schedule a second appointment for evaluation of their fracture: The first group will be scheduled for a second visit (standard treatment) as our daily practice after 1-3 months. They will be contacted after 2-6 months either by phone or email and will complete again some questionnaires (Quick DASH, satisfaction, return to work).
- Optional follow-up group: The alternative (Optional follow-up group) will be to take a handout describing the recovery and providing instructions for how to contact us should they get off course. The questionnaires will be repeated either by phone or email in 2-6 months.

SUMMARY:
Many common arm fractures have an excellent prognosis with little more than symptomatic treatment. When studying these fractures, investigators find that a substantial number of patients do not attend follow-up appointments. The difficulty of maneuvering in big cities, the cost of parking, the co-pay for the visit and the wait times for x-ray and doctor are all inconveniences that some patients might prefer to avoid. Building on prior research, it is appropriate to offer patients with common minor upper extremity fractures that have an excellent prognosis optional follow-up after the first visit. The plan would be to be available by phone, email and subsequent appointment at the patient's discretion if they felt that the recovery was off course. Benefit to individual participants is unlikely. The study will benefit the society as a whole, by providing a better understanding of these common fractures. It can also affect the economics of our health system by avoiding further follow-up appointments.

Primary null hypothesis: There is no difference in patient outcome 2-6 months after injury between patients that return for a second visit, and patients that do not.

Secondary null hypothesis: There is no difference in patient satisfaction 2-6 months after injury between patients that return for a second visit, and patients that do not.

DETAILED DESCRIPTION:
This study will employ a prospective, non-randomized design. After the questionnaires are filled the patients choose whether or not to schedule a second appointment for evaluation of their fracture: The first group will be scheduled for a second visit (standard treatment). The alternative (Optional follow-up) will be to take a handout describing the recovery and providing instructions for how to contact us should they get off course.

Since it is up to the subject to decide whether or not he or she wants a second appointment or the brochure, it is observational rather than interventional.

Evaluation: 2-6 months after injury all patients (independent of group) will be contacted by either phone or email by a blinded research assistant and asked to provide the following: pain with NRS (scale 0-10); three satisfaction questions; disability with use of Quick DASH; and if they returned to modified and regular work.

Patients in the standard group A will return to the Hand and Upper Extremity Service for their usual practice follow-up examination 1-3 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* adult (>18 years)
* English-speaking
* fracture with an excellent prognosis such as:
* nondisplaced mallet fracture
* stable, well-aligned metacarpal fracture
* all small finger metacarpal neck fractures
* non- or minimally displaced distal radius fracture treated in a removable splint
* isolated minimally displaced radial head fracture involving the radial neck or part of the articular surface

Exclusion Criteria:

* pregnant women
* no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult, English-speaking patients presenting to our outpatient clinic, that meet the inclusion criteria for this study will be invited to enroll at the time of the first visit at the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Disability with use of Quick DASH | Change from baseline at enrollment to follow-up at 2-6 months
  The Disabilities of Arm Shoulder and Hand (DASH) questionnaire is used frequently in hand and upper extremity research to assess disability. The Quick DASH is the short version of the DASH consisting of 11 questions.
  http://www.dash.iwh.on.ca/system/files/quickdash_questionnaire_2010.pdf

SECONDARY OUTCOMES:
Satisfaction | Change from baseline at enrollment to follow-up at 2-6 months
  The investigators measure the overall current patient satisfaction with an ordinal scale from 0 to 10, 0 being completely dissatisfied, 10 being completely satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: David Ring, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Hand Service, Department of Orthopaedic Surgery, Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Pike JM, Athwal GS, Faber KJ, King GJ. Radial head fractures--an update. J Hand Surg Am. 2009 Mar;34(3):557-65. doi: 10.1016/j.jhsa.2008.12.024. PMID 19258159
- [Background] Poolman RW, Goslings JC, Lee JB, Statius Muller M, Steller EP, Struijs PA. Conservative treatment for closed fifth (small finger) metacarpal neck fractures. Cochrane Database Syst Rev. 2005 Jul 20;2005(3):CD003210. doi: 10.1002/14651858.CD003210.pub3. PMID 16034891
- [Background] ten Berg PW, Ring D. Patients lost to follow-up after metacarpal fractures. J Hand Surg Am. 2012 Jan;37(1):42-6. doi: 10.1016/j.jhsa.2011.08.003. Epub 2011 Oct 19. PMID 22015075